CLINICAL TRIAL: NCT03837587
Title: Reliability, Validity of The Turkish Version of Craniofacial Pain and Disability Inventory
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Gazi University
Other Study IDs: 77082166-604.01.02-
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Validity; Reliability; Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Patients with temporomandibular disorders

SUMMARY:
This study, we are aim to make the Turkish version validity and reliability of the Cranifacial Pain and Disability Inventory, Jaw Functional Limitation Scale-20, and Jaw Functional Limitation Scale-8.

DETAILED DESCRIPTION:
Approximately 60% of individuals with temporomandibular disorders (TMD) reported increased pain intensity from midlevel to severe. This was seen at the end of the intervention or work related activities in the quarter of individuals. Therefore, the correct diagnosis of TMD is very important to reduce the economic cost. Craniofacial Pain and Disability Inventory (CF-PDI) is designed based on a biopsychosocial approach. Evidence has shown that CF-PDI is an well-structured, internal consistency, repeatable and valid, and that an objective outcome for the evaluation of pain and discomfort in patients with craniofacial pain. There is no Turkish version and validity study of CF-PDI. Each item is scored between 0-3. The total score ranged from 0 to 63, and a high score indicate a high level of discomfort. The aim of this study was to evaluate the validity and reliability of the Turkish version of CF-PDI. The study of validity and reliability is planned with 105 individuals with TMD. The sociodemographic characteristics of the individuals will be questioned by the investigators and then the patients will be evaluated with CF-PDI, Neck Disability Index (NDI), Tampa Scale for Kinesiophobia (TSK), Pain Catastrophizing Scale (PCS), Headache Impact Test-6 (HIT-6), Jaw Functional Limitation Scale (JFLS) (Turkish version) and Visual Analogue Scale (VAS). The test-retest will be re-administered by face-to-face interview technique after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Having a temporomandibular disorder
* Individuals who suited Temporomandibular Disorders/ Research Diagnostic Criteria classification

Exclusion Criteria:

* Pregnant,
* Canser,
* Trauma,
* Neurologic disorder,
* Infection,
* Trigeminal or postherpatic neuralgia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with temporomandibular disorders between the ages of 18-50
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Craniofacial Pain and Disability Inventory | 10 minutes
  Craniofacial Pain and Disability Inventory is a questionnaire that development to individuals with temporomandibular disorders. Each item is scored between 0-3. The total score range from 0 to 63, and a high score indicate a high level of discomfort. It is valid and reliable a questionnaire in clinic. Therefore, Turkish version must do.
Jaw Functional Limitation Scale-20 | 10 minutes
  Jaw Functional Limitation Scale-20 is a questionnaire that development to individuals with temporomandibular disorders. This questionnaire evaluates conditions of disability. Each item is scored between 0-10. It mean that "0= no limitation" and "10= severe limitation".The total score range from 0 to 200, and a high score indicate a high level of discomfort. It is valid and reliable a questionnaire in clinic. Therefore, Turkish version must do.
Jaw Functional Limitation Scale-8 | 5 minutes
  Jaw Functional Limitation Scale-8 is a questionnaire that development to individuals with temporomandibular disorders. This questionnaire evaluates conditions of disability. It is short form of Jaw Functional Limitation Scale-20. Each item is scored between 0-10. It mean that "0= no limitation" and "10= severe limitation".The total score range from 0 to 80, and a high score indicate a high level of discomfort. It is valid and reliable a questionnaire in clinic. Therefore, Turkish version must do.

CONTACTS AND LOCATIONS:
Overall Officials: Seyit ÇITAKER, Prof. Dr., Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Derived] Arikan H, Citaker S, Ucok C. Cross-cultural adaptation, reliability, and validity of the Turkish version of the Craniofacial Pain and Disability Inventory (CF-PDI/T) for individuals with temporomandibular disorders. Disabil Rehabil. 2023 Feb;45(3):523-533. doi: 10.1080/09638288.2022.2028909. Epub 2022 Feb 4. PMID 35119351